CLINICAL TRIAL: NCT03314233
Title: Delayed Cord Clamping for Intubation and Gentle Ventilation in Infants With Congenital Diaphragmatic Hernia
Brief Title: Delayed Cord Clamping for Congenital Diaphragmatic Hernia
Acronym: DING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-014125; K23HD084727 (NIH)
Record Dates: First submitted 2017-10-02; First posted 2017-10-19 (Actual); Results first posted 2019-12-10 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Intervention Model Description: Unblinded single-arm pilot interventional trial. All enrolled infants will receive the DING intervention (Delayed cord clamping for INtubation and Gentle ventilation)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DING intervention (Experimental): Delayed Cord Clamping
  Interventions: Procedure: DING

INTERVENTIONS:
Procedure: DING — Immediately after birth, the infant will be placed on a Lifestart trolley with an intact umbilical cord, intubated, and ventilated with the Children's Hospital of Philadelphia (CHOP) "gentle ventilation" protocol.

SUMMARY:
Congenital diaphragmatic hernia (CDH) is a congenital anomaly associated with a high risk of mortality and need for life-saving interventions such as extracorporeal membrane oxygenation (ECMO), nitric oxide, and vasopressor support. Although infants with CDH experience significant morbidity and mortality starting immediately after birth, high quality evidence informing delivery room resuscitation in this population is lacking.

Infants with CDH are at risk for pulmonary hypoplasia and pulmonary hypertension and often experience hypoxemia and acidosis during neonatal transition. The standard approach to DR resuscitation is immediate umbilical cord clamping (UCC) followed by intubation and mechanical ventilation. Animal models suggest that achieving lung aeration prior to UCC results in improved pulmonary blood flow and cardiac function compared with immediate UCC before lung aeration is established. Trials of preterm infants demonstrated that initiating respiratory support prior to UCC is safe and feasible. Because infants with CDH are at high risk for pulmonary hypertension and systemic hypotension, they may benefit from the hemodynamic effects of lung aeration before UCC, namely increased pulmonary blood flow, decreased pulmonary vascular resistance, and improved cardiac output. To date, this approach has not been studied in infants with CDH.

DETAILED DESCRIPTION:
Congenital diaphragmatic hernia (CDH) is a congenital anomaly associated with a high risk of mortality (29%) and need for life-saving interventions such as ECMO (33%), nitric oxide (62%), and vasopressor support (73%).1 Although infants with CDH experience significant morbidity and mortality starting immediately after birth, high quality evidence informing delivery room resuscitation in this population is lacking.

Infants with CDH are at risk for pulmonary hypoplasia and pulmonary hypertension and often experience hypoxemia and acidosis during neonatal transition. The standard approach to delivery room (DR) resuscitation is immediate UCC followed by intubation and mechanical ventilation. The goals of this strategy are to immediately recruit and aerate the lung for gas exchange and oxygenation, while simultaneously avoiding gaseous distention of the thoracic gastrointestinal contents.

Animal models suggest that achieving lung aeration prior to UCC results in improved pulmonary blood flow and cardiac function compared with immediate UCC before lung aeration is established. Trials of preterm infants demonstrated that initiating respiratory support prior to UCC is safe and feasible. Because infants with CDH are at high risk for pulmonary hypertension and systemic hypotension, they may benefit from the hemodynamic effects of lung aeration before UCC, namely increased pulmonary blood flow, decreased pulmonary vascular resistance, and improved cardiac output.

The investigators hypothesize that a sequence of intubation, gentle ventilation, and then umbilical cord clamping will result in improved cardiovascular transition after birth in infants with CDH. To date, this approach has not been studied in infants with CDH. The DING trial will assess the feasibility and safety of this intervention in infants with CDH.

ELIGIBILITY:
Inclusion Criteria:

1. Antenatal diagnosis of CDH, with care in the Center for Fetal Treatment
2. Gestational age ≥ 36 weeks at birth

Exclusion Criteria:

1. Multiple gestation
2. Major anomalies or aneuploidy
3. Enrolled in fetal endoluminal tracheal occlusion (FETO) trial
4. Palliative care planned or considered
5. Maternal diagnosis placenta previa, accreta, or abruption
6. Maternal diagnosis pre-eclampsia requiring Magnesium sulfate therapy at time of delivery
7. Obstetrics (OB) or Neonatal provider concerns for the clinical care of the mother or infant, or study team not available

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Foglia, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grover TR, Murthy K, Brozanski B, Gien J, Rintoul N, Keene S, Najaf T, Chicoine L, Porta N, Zaniletti I, Pallotto EK; Children's Hospitals Neonatal Consortium. Short-term outcomes and medical and surgical interventions in infants with congenital diaphragmatic hernia. Am J Perinatol. 2015 Sep;32(11):1038-44. doi: 10.1055/s-0035-1548729. Epub 2015 Mar 31. PMID 25825963

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DING Intervention
Started | 21 (21 mothers provided informed consent for participation in the trial.)
Completed | 20 (20 mothers who had provided informed consent met eligibility criteria at time of delivery.)
Not Completed | 1
Not completed — No longer eligible at time of delivery | 1

BASELINE CHARACTERISTICS:
Arm/Group | DING Intervention
Number analyzed (Participants) | 20
Age, Customized [Mean (Standard Deviation); unit: weeks]
  Gestational Age | 38.7 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Infants Who Are Intubated Prior to Umbilical Cord Clamping
Description: Infants who are intubated and have ventilation initiated prior to umbilical cord clamping
Time Frame: 3 minutes of life
Measure: Count of Participants; unit: Participants
Arm/Group | DING Intervention
Number analyzed (Participants) | 20
Participants | 17

2. Secondary Outcome: Mean Arterial Potential of Hydrogen (pH) in Arterial Blood
Description: Arterial pH on first blood gas
Time Frame: Approximately 1 hour of life
Population: 1 of the 20 infants randomized to the intervention was diagnosis with a second major anomaly postnatally and was not included in the secondary outcome results.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | DING Intervention
Number analyzed (Participants) | 19
pH | 7.02 (0.15)

3. Secondary Outcome: Mean Partial Pressure of O2 in Arterial Blood (PaO2)
Description: Arterial PaO2 on first blood gas
Time Frame: Approximately 1 hour of life
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: PaO2
Arm/Group | DING Intervention
Number analyzed (Participants) | 19
PaO2 | 47 [39 to 52]

4. Secondary Outcome: Oxygenation Index (OI)
Description: Oxygenation index [OI] with first obtained blood gas
Time Frame: First obtained blood gas
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: oxygenation index
Arm/Group | DING Intervention
Number analyzed (Participants) | 19
oxygenation index | 17.5 [12.8 to 25.5]

5. Secondary Outcome: Proportion of Infants Who Require Vasopressors
Description: Proportion of infants who require vasopressors in first 48 hours of life
Time Frame: First 48 hours of life
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | DING Intervention
Number analyzed (Participants) | 19
Participants | 13

6. Secondary Outcome: Presence of Severe Pulmonary Hypertension
Description: Presence of severe pulmonary hypertension on first echocardiogram
Time Frame: Approximately 24 hours of life
Population: 1 of the 20 infants randomized to the intervention was diagnosis with a second major anomaly postnatally and was not included in the secondary outcome results. 1 trial participant was supported with ECMO when the echocardiogram was obtained and therefore was not assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | DING Intervention
Number analyzed (Participants) | 18
Participants | 12

7. Secondary Outcome: Proportion of Infants Who Require Extracorporeal Membrane Oxygenation (ECMO) Treatment
Description: Proportion of infants who require ECMO treatment in first 7 days of life
Time Frame: 7 days of life
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | DING Intervention
Number analyzed (Participants) | 19
Participants | 7

8. Secondary Outcome: Mortality in First 7 Days of Life
Description: Proportion of infants with mortality in the first 7 days of life
Time Frame: First 7 days of life
Measure: Count of Participants; unit: Participants
Arm/Group | DING Intervention
Number analyzed (Participants) | 20
Participants | 0

ADVERSE EVENTS:
Time Frame: 24 hours following allocation to the DING intervention.
Arm/Group | DING Intervention
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DING Intervention (N=20)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT03314233/Prot_SAP_000.pdf